CLINICAL TRIAL: NCT02051686
Title: Hemostasis in Open Acetabulum and Pelvic Ring Surgery Using Tranexamic Acid: A Prospective, Randomized, Controlled Study
Brief Title: Hemostasis in Open Acetabulum and Pelvic Ring Surgery Using Tranexamic Acid
Acronym: TXA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Brett Crist, Assistant Professor, Co-Director of Trauma Services, Co-Director Orthopaedic Trauma Fellowship, Department of Orthopaedic Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1208444
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-01

CONDITIONS: Acetabulum Fractures
Keywords: Acetabulum Fractures; Pelvic Ring Injuries; Tranexamic Acid
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic Acid (Active Comparator): Group I will receive 10 mg/kg TXA loading dose approximately 15 minutes before surgical start time and then 1 mg/kg/h TXA infusion over 10 hours.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): The control group will receive a similar volume load of normal saline and maintenance doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — 10 mg/kg TXA loading dose approximately 15 minutes before surgical start time and then 1 mg/kg/h TXA infusion over 10 hours.
  Other Names: Cyklokapron; Transamin
  Arms: Tranexamic Acid
Drug: Placebo — The control group will receive a similar volume load of normal saline and maintenance doses.
  Arms: Placebo

SUMMARY:
This study is investigating the use of tranexamic acid (TXA) in patients with pelvis and/or hip socket fractures that require surgery. TXA is FDA-approved in patients with hemophilia for short-term use to reduce hemorrhage and the need for replacement blood during tooth extraction. However, it has also been used extensively in severely injured patients after major trauma and during elective hip and knee replacements. Previous studies indicate TXA may reduce blood loss and the need for blood transfusions while being safe for use in most patients. TXA is fairly inexpensive and easy to obtain.

The purpose of this study is to determine if TXA will make surgery in patients with pelvis and/or hip socket fractures safer and more cost efficient.

DETAILED DESCRIPTION:
Study candidates will be identified as they present to the University Hospital emergency room and will be recruited for enrollment. Randomization will occur by electronic randomization software. Prior to surgery, the pharmacy will be notified of an enrolled patient and will be responsible for randomization and creating either a placebo intravenous dose or a treatment study dose. Both study groups will receive the standard of care treatment for intra-operative hemorrhage control.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age or greater) with acetabulum fractures and/or pelvic ring injuries that require operative fixation via an open surgical approach

Exclusion Criteria:

* Revision surgery
* Surgery occurring more than 2 weeks post-injury
* History of blood dyscrasia or renal insufficiency
* History of any thromboembolic disease
* Pregnancy or nursing, color vision defects
* History of retinal detachment/degeneration
* Intracranial hemorrhage
* Hypersensitivity to tranexamic acid
* Contraceptive Use (estrogens/progestins)
* FEIBA (anti-inhibitor coagulant complex) use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett D Crist, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tranexamic Acid | Placebo
Started | 42 | 46
Completed | 42 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tranexamic Acid: Patients in the intervention group were administered a 10mg/kg preoperative dose of tranexamic acid within 30 minutes prior to surgery followed by a 10mg/kg infusion over a 4hr period during surgery.
- Placebo: Patients in the control group received an equal volume and rate of normal saline.
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Placebo | Total
Number analyzed (Participants) | 42 | 46 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (15.6) | 39.7 (16.1) | 40.7 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 31 | 34 | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 46 | 88

OUTCOME MEASURES:

1. Primary Outcome: Intra-operative Blood Loss
Time Frame: Day of Surgery
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 42 | 46
Milliliters | 727.6 (702.52) | 560.1 (378.4)

2. Secondary Outcome: Number of Participants That Required an Allogenic Transfusion
Time Frame: Perioperative (hospitalized period)
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 42 | 46
Participants | 21 | 15

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Tranexamic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/46
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/46
Other Adverse Events (participants affected / at risk) | 0/42 | 0/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid (N=42) | Placebo (N=46)
Venous thromboembolism (Blood and lymphatic system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes